CLINICAL TRIAL: NCT01128335
Title: A 24-month Randomized Multicenter Study Evaluating Efficacy, Safety, Tolerability and Pharmacokinetics of Sotrastaurin and Tacrolimus vs. a Tacrolimus/Mycophenolate Mofetil-based Control Regimen in de Novo Liver Transplant Recipients
Brief Title: Efficacy, Safety, Tolerability, Pharmacokinetics of Sotrastaurin-tacrolimus vs. Mycophenolic Acid-tacrolimus in de Novo Liver Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAEB071B2201; 2007-001776-36
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2016-11

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation; HCV-negative recipient; deceased donor; sotrastaurin; oran transplantation; tacrolimus
MeSH Terms: interventions — BID protein, human; Tacrolimus; sotrastaurin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Arm 1 (Active Comparator): MMF(1000mg bid) + tacrolimus + standard of care medications
  Interventions: Drug: MMF(1000mg bid) + tacrolimus + standard of care medications
- Arm 2 (Experimental): sotrastaurin (200mg bid) + tacrolimus + standard of care medications
  Interventions: Drug: sotrastaurin (200mg bid) + tacrolimus + standard of care medications
- Arm 3 (Experimental): sotrastaurin (200mg bid) + tacrolimus + standard of care medications
  Interventions: Drug: sotrastaurin (200mg bid) + tacrolimus + standard of care medications
- Arm 4 (Experimental): sotrastaurin (300 mg bid) + tacrolimus + standard of care medications
  Interventions: Drug: sotrastaurin (300 mg bid) + tacrolimus + standard of care medications

INTERVENTIONS:
Drug: MMF(1000mg bid) + tacrolimus + standard of care medications — MMF(1000mg bid) + tacrolimus + standard of care medications
  Arms: Arm 1
Drug: sotrastaurin (200mg bid) + tacrolimus + standard of care medications — sotrastaurin (200mg bid) + tacrolimus + standard of care medications
  Arms: Arm 2
Drug: sotrastaurin (200mg bid) + tacrolimus + standard of care medications — sotrastaurin (200mg bid) + tacrolimus + standard of care medications
  Arms: Arm 3
Drug: sotrastaurin (300 mg bid) + tacrolimus + standard of care medications — sotrastaurin (300 mg bid) + tacrolimus + standard of care medications
  Arms: Arm 4

SUMMARY:
This study will assess the safety and efficacy of different doses of sotrastaurin when combined with tacrolimus for the prevention of acute rejection after de novo liver transplantation.

ELIGIBILITY:
Inclusion criteria:

* Recipients of any race, 18 years or older
* Recipients of primary de novo orthotopic liver transplant from a deceased donor
* Recipients of a kidney with a cold ischemia time < 30 hours
* HCV-negative recipients

Exclusion criteria:

* Prior organ/cellular transplant or multiple organ transplant
* MELD-score > 35
* HCC > Milan criteria
* Donor age < 12 years
* Cold ischemia > 15 hours
* Patients who are treated with drugs that are strong inducers or inhibitors of cytochrome P450 3A4 (CYP3A4) or drugs with QT-prolonging properties

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of primary efficacy failure defined as composite efficacy endpoint (treated BPAR of Banff grade ≥ 1, graft loss, or death) in the different treatment arms. | Month 6

SECONDARY OUTCOMES:
Evaluate renal allograft function post-transplantation (estimated GFR by MDRD equation; estimated creatinine clearance by Cockcroft-Gault formula; serum creatinine). | Months 3, 6, 12, and 24
Occurrence of primary efficacy failure defined as composite efficacy endpoint (treated BPAR of Banff grade ≥ 1, graft loss, or death) in the different treatment arms. | Months 12, 24
Occurrence of rejection requiring T-cell depleting antibody, occurrence of treated biopsy-proven acute rejections of Banff grade ≥ 1 that is steroid-resistant | Months 6, 12, 24
Safety and tolerability ((serious) adverse events (specifically: gastrointestinal AEs and cardiac AEs, serious infections), laboratory abnormalities, vital signs, electrocardiograms, physical examination). | Months 3, 6, 12, 24

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmceuticals, Study Director — Novartis Pharmaceuticals
Locations (38):
- United States (8):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, San Martín, Buenos Aires
- Austria (2):
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, London, Ontario, Canada
- Czechia (2):
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Brno
- Novartis Investigative Site, HUS, Finland
- France (6):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Villejuif
- Germany (6):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Regensburg
- Italy (3):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
- Spain (4):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Valencia, Valencia
- Novartis Investigative Site, Zurich, Switzerland

REFERENCES:
- [Result] Pascher A, De Simone P, Pratschke J, Salame E, Pirenne J, Isoneimi H, Bijarnia M, Krishnan I, Klupp J. Protein kinase C inhibitor sotrastaurin in de novo liver transplant recipients: a randomized phase II trial. Am J Transplant. 2015 May;15(5):1283-92. doi: 10.1111/ajt.13175. Epub 2015 Feb 12. PMID 25677074
- See also: Results for CAEB071B2201 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8843